CLINICAL TRIAL: NCT01367678
Title: Directly Measured Mucosal Pressure for Two Different Extraglottic Airway Devices
Brief Title: Mucosal Pressure of the Laryngeal Mask Airway Supreme Versus the i-Gel in Paralyzed Anesthetized Female Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, ChristianKeller, MD, M.Sc., Schulthess Klinik
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Schulthess_Anä_1
Record Dates: First submitted 2011-06-03; First posted 2011-06-07 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Device Induced Injury; Necrosis, Pressure; Complication of Device Insertion; Airway Morbidity
MeSH Terms: conditions — Necrosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laryngeal Mask Airway Supreme (Experimental): Directly measured mucosal pressures
  Interventions: Device: Laryngeal Mask Airway Supreme
- i-Gel (Experimental): Directly measured mucosal pressures
  Interventions: Device: i-Gel extraglottic airway device

INTERVENTIONS:
Device: Laryngeal Mask Airway Supreme — Directly measured mucosal pressures
  Other Names: Supreme
  Arms: Laryngeal Mask Airway Supreme
Device: i-Gel extraglottic airway device — Directly measured mucosal pressures
  Other Names: i-Gel
  Arms: i-Gel

SUMMARY:
In the following randomized non-crossover study, the investigators test the hypothesis that directly measured mucosal pressure differ between the laryngeal mask airway (LMA) Supreme and the i-Gel in paralyzed anesthetized females.

Thirty females aged 19-65 years were randomly allocated to receive either the size 4 LMA Supreme or i-Gel for airway management. Microchip sensors were attached to the LMA Supreme/i-Gel at four locations corresponding to the A, base of tongue; B, distal oropharynx; C, hypopharynx; and D, pyriform fossa.

Insertion success rate and oropharyngeal leak pressure were also measured.

ELIGIBILITY:
Inclusion Criteria:

* ASA I/II
* female
* age 19-65 years

Exclusion Criteria:

* < 19 years
* had a known or predicted difficult airway
* a body mass index > 35 kg m-2, or
* were at risk of aspiration

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
pharyngeal mucosal pressure | every 5 minutes during steady state anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Christian Keller, MD, M.Sc., Study Director — Schulthess Klinik
Locations (2):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria
- Christian Keller MD, M.Sc., Zurich, Switzerland